CLINICAL TRIAL: NCT05332912
Title: Assessing the Malleability of Spatial Abilities in Individuals With Down Syndrome
Brief Title: Assessing Malleability of Spatial Abilities in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Ed Merrill, Professor Emeritus, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-08-2644
Record Dates: First submitted 2022-04-02; First posted 2022-04-18 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Typically developing children will be compared to adolescents/young adults with Down syndrome (groups matched on non-verbal ability).
  A delayed start condition (verbal experience instead of spatial ability experience) of eight weeks will be used for 1/2 of participants in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Participants will receive 16 weeks of spatial ability experience.
  Interventions: Behavioral: Spatial Ability Experience
- Delayed (Placebo Comparator): Participants will receive 8 weeks of verbal ability experience prior to receiving 8 weeks of spatial ability experience.
  Interventions: Behavioral: Spatial Ability Experience

INTERVENTIONS:
Behavioral: Spatial Ability Experience — Participants will engage in puzzle construction, block play, visual search, hide and seek

SUMMARY:
Based on available literature and our own preliminary research, the researchers have concluded that persons with Down syndrome (DS) exhibit difficulties in utilizing the specific spatial abilities of mental rotation and perspective taking and performing complex spatial tasks such as wayfinding and environmental learning. A weakness in spatial abilities may have many direct applications to daily life, ranging from activities such as tying shoes to using hand tools and navigating the environment. Spatial abilities also serve as a cognitive foundation for many other complex skills such as solving mathematical problems and using spatial language for giving and receiving directions. Moreover, spatial abilities are used in a variety of specialty jobs such as grocery stocking, packaging, and assembling, which are among the most commonly reported jobs for adults with DS. Hence, a new focus on spatial ability and its modifiability in persons with DS is clearly warranted. The primary goal of the research proposed in this application is to evaluate the malleability of mental rotation and perspective taking in people with DS through providing intentional experience with numerous spatial activities. Two groups of participants will be tested over the course of the project: adolescents and young adults with DS and typically developing (TD) children. Following an initial evaluation of performance on the two abilities, participants will receive up to eight sessions of spatial activity experience utilizing puzzle construction, block building, and computer search tasks. Following the experience sessions, spatial abilities of participants will be re-evaluated. These data will be used to investigate two specific aims. First, the researchers investigate whether spatial abilities of persons with DS can be modified by experience with spatial activities. Second, the researchers investigate whether the degree of modification observed for persons with DS can reduce performance differences between them and TD children. The researchers also consider whether performance on the PPVT, Raven's matrices, and Chronological Age are associated with any benefits from spatial ability experience.

DETAILED DESCRIPTION:
Participants will take part in a study designed to facilitate the development of two spatial abilities: Mental Rotation and Visual Perspective Taking. Mental rotation reflects the ability to mentally manipulate a small object without physically rotating it. Perspective taking reflects the ability to imagine what a large environment would look like from a different position. Both abilities are important for engaging in everyday spatial activities such as navigating the environment without getting lost. The researchers have constructed four tasks to provide experience with these two abilities over the course of approximately four months. There will be an initial assessment (one week), followed by eight weeks of experiences using four different spatial ability games, a second assessment, eight more weeks of experience, and then a third assessment.

The initial assessment will include four measures:

Ravens 2 Matrices: The Ravens 2 Matrices is a 60 item measure of nonverbal ability. The subtest measures a participant's ability to solve problems, identify relationships, and complete visual analogies without testing language skill. The examiner shows the participant pictures or abstract designs that follow a pattern, with one element missing. The participant is instructed to point to a picture that will complete the pattern. Participants will be matched on raw score performance. Completing the subtest should take less than 15 minutes for most participants. We will use Age-Equivalent scores as our measure of performance. The score can range from 48 to 239 months and are standardized scores reflecting participant's ability level at the time of testing.

PPVT-4: The PPVT - 4 is a norm-referenced test for measuring receptive vocabulary of children and adults. The test is administered individually. Each item consists of four colored pictures that serve as response choices on each page. For each item, the examiner says a word and the examinee selects the picture option that best represents the word's meaning. The test is normed for 2 years, 6 months to 90 years. Average time to administer the test is 10 - 15 minutes. We will use Age-Equivalents scores for the PPVT. Age-equivalent scores can range from 30 to 218 months and are standardized scores.

Mental Rotation Assessment - On each trial, participants will be presented a shape (e.g., a block letter L) in the center of a computer screen that completes one of two silhouettes presented in rectangles at the bottom of the same screen. The open area in one rectangle is the mirror image of the open area in the second rectangle. The shape in the center of the screen will fit one of the rectangles when horizontal. The shape can be rotated from horizontal by 0, 45, 90, 135, 180, 225, 270, or 315 degrees. Participants respond by touching the rectangle into which the shape will fit once oriented properly (using touchscreen technology).

Number of correct responses (excluding 0 rotation trials) are counted. Scores can range from 0 to 18. To directly compare performance on Motel Rotation with performance on Perspective Taking, percent of total available points are used on the analyses.

Perspective Taking - Participants will be seated at a table with four chairs and four different objects (e.g., street lamp, mailbox, stop sign, traffic signal) representing each location on the corner of a city block in front of each chair. A stuffed animal is placed behind each object. One experimenter walks around the table stopping at various locations around the table (12 different locations). At each location, the participant is told that the experimenter is taking a picture from that location and he/she is asked to look at four pictures. The task is to select the picture that the experimenter has just taken. The four pictures consist of the participant's point of view, a mirror image of the participant's point of view, the experimenter's (correct) point of view, and a mirror image of the experimenter's point of view. This task will take 5 - 10 minutes. Participants are given 3 points for selecting the experimenter's (correct) perspective, 2 points for selecting the mirror image of the experimenter's perspective, 1 point for selecting the view opposite their own perspective, and 0 points for selecting their own perspective. Total points in this task could range from 0 to 36.

Percent of total available points earned on this task is used as the measure of perspective taking to allow comparison with mental rotation performance.

Assessments 2 and 3 will include only Mental Rotation and Perspective Taking Assessments.

Spatial Ability Experience will include two tasks of Object manipulation and two Large Environment Experiences.

Object Manipulation Experience: Two categories of tasks will be used to provide object manipulation experience: LEGO Block Play and Puzzle Construction. One task will be used in each spatial ability experience, with tasks alternating between sessions.

LEGO Block Play: Participants and experimenter will each have 20 multi-colored and multi-shaped connecting blocks. During play, the participant and experimenter will alternate creating structures and copying what the other has created during the 15-minute interval. No specific corrective feedback will be given during the experience, although participants will be asked if the construction matches the model. Object manipulation rather than accuracy is the basis of the experience. Participants will be allowed to take as long as needed to complete their copy of each structure.

Puzzle Construction: The researchers will select puzzles that include 4, 8, 12, 16, or 20 puzzle pieces. All puzzles will have pieces that need to be rotated to fit the puzzle board to provide the necessary object manipulation experience. The puzzle board will also include the outline of the shapes of the pieces. Hence, participants will need to match the outline of the piece with the rotated actual piece to efficiently complete the puzzle. Touching each piece with a finger will rotate the piece and removing the finger will stop the rotation. Participants will be given five puzzles to complete during the experience session. The participant will be given 3 minutes to complete each puzzle. If the participant completes the puzzle, the next larger size puzzle will be used for the participant's next opportunity. If the participant fails to complete the puzzle, the size of the puzzle will be reduced by one level.

Large Environment Experience: Two categories of tasks using a large-scale virtual environment will be used to provide object manipulation experience: Hide and Seek and Wayfinding. One task will be used in each spatial ability experience, with tasks alternating between sessions.

Hide and Seek Video Game: Several settings are used to limit boredom with the task. For example, participants are shown a panoramic view in a living room. In the center of the picture is a stuffed animal who was identified as the seeker in the game. They are then shown a view of what the seeker could see - which includes four different color boxes. They are told another animal (e.g., dog) is hiding behind one of the boxes. Then they are shown what the dog could see looking back at the seeker. They are asked to identify where the dog is hiding based on what the dog could see. If incorrect, they are asked to try again. They are given four different animals to located during each session the task is used.

Wayfinding Video Game: Children will be exposed to a scene using Google street view and asked to search for specific targets that can be scene along the path. In order to complete the task, the participant will need to be able to identify the targets from different perspectives.

Children who are assigned to the Control condition will receive the spatial ability experiences following an eight-week delay after the initial assessment.

ELIGIBILITY:
Inclusion Criteria:

* Typically Developing Children ages 4.0 years to 9.0 years
* Individuals with Down Syndrome ages 10.0 - 25.0
* Verbal Comprehension Ability at 4.0 years or above

Exclusion Criteria:

* Inability to follow verbal instructions
* Inability of use tablet computer

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward C Merrill, Phd, Principal Investigator — University of Alabama, Tuscaloosa
Locations (1):
- University of Alabama, Tuscaloosa, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be available upon request after the study is completed, data has been analyzed, and the primary data has been published or within 5 years of study completion if data has not been published. Requests can be made to the PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following publication of the primary data or within 5 years of study completion if data has not been published. Data will be available for a minimum of 5 years.
Access Criteria: Requests will be accepted from behavioral researchers with a PhD or equivalent who identify a specific purpose and research appropriate justification for accessing the IPD. Requests will be reviewed by the PI and the sub-contract PI.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants self-identified to the researchers by responding to notices placed in various locations, including daycare centers, Children helping science website, Down syndrome organizations (locally and nation-wide), etc. Following contact that included providing details of the project, potential participants who met criteria were sent informed consent documents. Those who returned signed consent documents were identified as enrolled in the study. Dates:
Pre-assignment Details: Treatment vs delayed treatment (control) were identified in waves (as control required matching with the treatment group on nonverbal ability). CoVid restrictions at the start of the study and use of remote only testing impacted recruit of individuals with Down syndrome. Hence, all participants with Down Syndrome were assigned to a treatment group to maximize their contribution to the research. Typically developing children served as controls for both groups.
Groups:
- Typically Developing Children Immediate Intervention: Children Participants received 16 weeks of spatial ability experience.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Typically Developing Children Delayed Intervention: Children Participants received 8 weeks of spatial ability experience that was initiated eight weeks following the initial assessment (no intervening task) and immediately following the second assessment.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Down Syndrome Participants Immediate Intervention: Down Syndrome Participants received 16 weeks of spatial ability experience.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Down Syndrome Participants Deleayed Intervention: Down Syndrome Participants received 8 weeks of spatial ability experience that was initiated eight weeks following the initial assessment (no intervening task) and immediately following the second assessment.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play,
Period: Overall Study
Arm/Group | Typically Developing Children Immediate Intervention | Typically Developing Children Delayed Intervention | Down Syndrome Participants Immediate Intervention | Down Syndrome Participants Deleayed Intervention
Started | 30 | 24 | 30 | 0
Completed | 30 | 23 | 27 | 0
Not Completed | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The difficulty of recruiting Down Syndrome participants during the CoVid period coupled with parents' reluctance to participate in a long-term study that might not provide maximum benefit to their own child led us to prioritize completing the Immediate Intervention condition for Down Syndrome participants to yield results with maximum overall utility. Hence, no Down Syndrome individuals were assigned to the Delayed Intervention condition.
Groups:
- Typically Developing Children Immediate Intervention: Children Participants will receive 16 weeks of spatial ability experience.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Typically Developing Children Delayed Intervention: Children Participants will receive 8 weeks of verbal ability experience prior to receiving 8 weeks of spatial ability experience.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Down Syndrome Participants Immediate Intervention: Down Syndrome Participants will receive 16 weeks of spatial ability experience.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Down Syndrome Participants Delayed Intervention: Down Syndrome Participants will receive 8 weeks of verbal ability experience prior to receiving 8 weeks of spatial ability experience.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Total: Total of all reporting groups
Arm/Group | Typically Developing Children Immediate Intervention | Typically Developing Children Delayed Intervention | Down Syndrome Participants Immediate Intervention | Down Syndrome Participants Delayed Intervention | Total
Number analyzed (Participants) | 30 | 24 | 30 | 0 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 24 | 16 |  | 70
  Between 18 and 65 years | 0 | 0 | 14 |  | 14
  >=65 years | 0 | 0 | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 15 |  | 42
  Male | 13 | 14 | 15 |  | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 5 |  | 15
  Not Hispanic or Latino | 24 | 20 | 25 |  | 69
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 3 | 2 | 2 |  | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 6 | 4 | 4 |  | 14
  White | 21 | 18 | 24 |  | 63
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 24 | 30 |  | 84
Ravens Progressive Matrices 2nd Edition [Mean (Standard Deviation); unit: Performance Age Equivalence in Months] — We used Age-Equivalent scores as our measure of performance. The score can range from 48 to 239 months. The score reflects the average age at which a specific aptitude score is typically achieved.
  Performance Age Equivalence in Months | 109 (39) | 90 (30) | 83 (35) |  | 94 (36)
Peabody Picture Vocabulary Test 4th Edition [Mean (Standard Deviation); unit: Performance Age Equivalence in Months] — We used Age Equivalence scores for the measure of performance (reported in months). The score can range from 30 to 218 months. This measure reflects the average age at which a specific aptitude score is obtained.
  Performance Age Equivalence in Months | 121 (50) | 105 (37) | 93 (24) |  | 107 (41)
Mental Rotation Ability [Mean (Standard Deviation); unit: Number Correct out of 18] — Number of times participants selected the correct rotated response on 18 trials. Range of scores is 0 - 18. A score of 9 would reflect chance level performance.
  Number Correct out of 18 | 15.4 (2.5) | 14.5 (3.7) | 13.3 (4.1) |  | 14.4 (4)
Visual Perspective Taking Ability [Mean (Standard Deviation); unit: Number of Total Points out of 24] — Participants received 8 trials in which they judged another's point of view. They received 3 points for choosing the correct point of view, 2 points for the point of view opposite the correct one, and 1 point for choosing a view not their own. The receive 0 points if they chose their own point of view. Range of scores 0 to 24. Chance performance would be 12 (an average of 1.5 points per trial).
  Number of Total Points out of 24 | 15.9 (6.5) | 13.6 (6.6) | 11.5 (4.5) |  | 13.7 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mental Rotation Ability at 8 Weeks
Description: The Mental Rotation Assessment was used to assess ability to match objects rotated at varying degrees from a standard. Number of correct matches out of 18 possible matches over all rotations (excluding 0 degrees) was used as a measure of performance. Minimum score = 0. Maximum score = 18. Higher scores reflect better performance. Change in Mental Rotation Ability was calculated by subtracting Baseline (Time 1) Assessment scores from 8 Week (Time 2) Assessment scores.
Time Frame: Following 8 weeks of experience training.
Population: No Down Syndrome participants took part in the Delayed Intervention Condition.
Measure: Mean (Standard Deviation); unit: Amount of Change in Number Correct Items
Groups:
- Typically Developing Children Delayed Intervention: Children Participants received 8 weeks of spatial ability experience. Experience training was initiated eight weeks following the initial assessment (no intervening task) and immediately following the second assessment.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Down Syndrome Participants Delayed Intervention: Down Syndrome participants received 8 weeks of spatial ability experience. Experience training was initiated eight weeks following the initial assessment (no intervening task) and immediately following the second assessment.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
Arm/Group | Typically Developing Children Immediate Intervention | Typically Developing Children Delayed Intervention | Down Syndrome Participants Immediate Intervention | Down Syndrome Participants Delayed Intervention
Number analyzed (Participants) | 30 | 23 | 27 | 0
Amount of Change in Number Correct Items | 0.0 (0.8) | -0.6 (3.3) | .82 (2.8) |
Statistical Analysis 1: Comparison: Down Syndrome Participants Immediate Intervention; Null Hypothesis: Participants with Down Syndrome will exhibit no change in number of correct items in Mental Rotation performance following 8 weeks of experiential training; Test type: Superiority; p = .066, t-test, 1 sided; df = 26
Statistical Analysis 2: Comparison: Typically Developing Children Delayed Intervention vs Down Syndrome Participants Immediate Intervention; Null Hypothesis: Amount of change in Mental Rotation performance following 8 weeks of experiential training will not differ for participants with Down Syndrome who received 8 weeks of experiential intervention and Typically Developing Children in the Delayed Intervention who had not received 8 weeks of intervention; Test type: Superiority; p = .056, t-test, 1 sided
Statistical Analysis 3: Comparison: Typically Developing Children Immediate Intervention vs Down Syndrome Participants Immediate Intervention; Null Hypothesis: Amount of change in Mental Rotation performance following 8 weeks of experiential training will not differ for Typically Developing Children Immediate Intervention and Down Syndrome Participants Immediate intervention; Test type: Superiority; p = .65, t-test, 2 sided; df = 55

2. Primary Outcome: Change in Mental Rotation Ability at 16 Weeks
Description: The Mental Rotation Assessment was used to assess ability to match objects rotated at varying degrees from a standard. Number of correct matches out of 18 possible matches over all rotations (excluding 0 degrees) was used as a measure of performance. Minimum score = 0. Maximum score = 18. Higher scores reflect better performance. Change in Mental Rotation Ability was calculated by subtracting Baseline (Time 1) Assessment scores from 8 Week (Time 3) Assessment scores.
Time Frame: Following 16 weeks of experience training.
Population: No Down Syndrome participants took part in the Delayed Intervention Condition.
Measure: Mean (Standard Deviation); unit: Amount of Change in Number Correct Items
Groups:
- Typically Developing Children Delayed Intervention; Down Syndrome Participants Delayed Intervention: Participants received 8 weeks of spatial ability experience. Experience training was initiated eight weeks following the initial assessment (no intervening task) and immediately following the second assessment.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
Arm/Group | Typically Developing Children Immediate Intervention | Typically Developing Children Delayed Intervention | Down Syndrome Participants Immediate Intervention | Down Syndrome Participants Delayed Intervention
Number analyzed (Participants) | 30 | 23 | 27 | 0
Amount of Change in Number Correct Items | 1.3 (2.3) | 1.0 (2.2) | 0.8 (2.9) |
Statistical Analysis 1: Comparison: Down Syndrome Participants Immediate Intervention; Null Hypothesis: Participants with Down Syndrome will exhibit no change in number of correct items in Mental Rotation performance following 16 weeks of experiential training; Test type: Superiority; p = .039, t-test, 1 sided
Statistical Analysis 2: Comparison: Typically Developing Children Delayed Intervention vs Down Syndrome Participants Delayed Intervention; Null Hypothesis: Participants with Down Syndrome in the Immediate Intervention condition and received 16 weeks of experiential training in Mental Rotation will exhibit a similar change in performance as Typically Developing Children in the Delayed Intervention condition who received only 8 weeks of experiential training; Test type: Superiority; p = .32, t-test, 2 sided; df = 48
Statistical Analysis 3: Comparison: Typically Developing Children Immediate Intervention vs Down Syndrome Participants Immediate Intervention; Null Hypothesis: Amount of change in Mental Rotation performance following 16 weeks of experiential training will not differ for Typically Developing Children Immediate Intervention and Down Syndrome Participants Immediate intervention; Test type: Superiority; p = .73, t-test, 2 sided — df = 55

3. Primary Outcome: Change in Perspective Taking Ability at 8 Weeks
Description: Measure Description: Participants received 8 trials in which they judged another's point of view. Scores could range from 0 to 24. . Change in Perspective Taking Ability was calculated by subtracting Baseline (Time 1) Assessment scores from 8 Week (Time 2) Assessment scores.
Time Frame: Following 8 weeks of experience training.
Population: No Down Syndrome participants took part in the Delayed Intervention Condition.
Measure: Mean (Standard Deviation); unit: Change in Performance Points Awarded
Arm/Group | Typically Developing Children Immediate Intervention | Typically Developing Children Delayed Intervention | Down Syndrome Participants Immediate Intervention | Down Syndrome Participants Delayed Intervention
Number analyzed (Participants) | 30 | 23 | 27 | 0
Change in Performance Points Awarded | 0.9 (3.1) | 2.5 (4.1) | 1.6 (4.0) |
Statistical Analysis 1: Comparison: Down Syndrome Participants Immediate Intervention; Null Hypothesis: Participants with Down Syndrome will exhibit no change in Perspective Taking performance following 8 weeks of experiential training; Test type: Superiority; p = .023, t-test, 1 sided; df = 26
Statistical Analysis 2: Comparison: Typically Developing Children Delayed Intervention vs Down Syndrome Participants Immediate Intervention; Null Hypothesis: Amount of change in Perspective Taking performance following 8 weeks of experiential training will not differ for participants with Down Syndrome who received 8 weeks of experiential intervention and Typically Developing Children in the Delayed Intervention who had not received 8 weeks of intervention; Test type: Superiority; p = .23, t-test, 1 sided; df = 48
Statistical Analysis 3: Comparison: Typically Developing Children Immediate Intervention vs Down Syndrome Participants Immediate Intervention; Null Hypothesis: Amount of change in Mental Rotation will not differ for participants with Down Syndrome in the Immediate Intervention Condition who received 8 weeks of experiential intervention and Typically Developing Children in the Immediate Intervention who also received 8 weeks of intervention; Test type: Superiority; p = .42, t-test, 2 sided; df = 55

4. Primary Outcome: Change in Perspective Taking Ability at 16 Weeks
Description: Participants received 8 trials in which they judged another's point of view. Scores could range from 0 to 24. Change in Perspective Taking Ability was calculated by subtracting Baseline (Time 1) Assessment scores from 16 Week (Time 3) Assessment scores.
Time Frame: Following 16 weeks of experience training.
Population: No Down Syndrome participants took part in the Delayed Intervention Condition.
Measure: Mean (Standard Deviation); unit: Change in Performance Points Awarded
Arm/Group | Typically Developing Children Immediate Intervention | Typically Developing Children Delayed Intervention | Down Syndrome Participants Immediate Intervention | Down Syndrome Participants Delayed Intervention
Number analyzed (Participants) | 30 | 23 | 27 | 0
Change in Performance Points Awarded | 1.0 (3.7) | 1.6 (5.1) | 2.4 (5.1) |
Statistical Analysis 1: Comparison: Down Syndrome Participants Immediate Intervention; Null Hypothesis: Participants with Down Syndrome will exhibit no change in Perspective Taking performance following 16 weeks of experiential training; Test type: Superiority; p = .01, t-test, 1 sided; df = 26
Statistical Analysis 2: Comparison: Typically Developing Children Delayed Intervention vs Down Syndrome Participants Delayed Intervention; Null Hypothesis: Amount of change in Perspective Taking will not differ for participants with Down Syndrome in the Immediate Intervention Condition who received16 weeks of experiential intervention and Typically Developing Children in the Delayed Intervention condition who received 8 weeks of intervention; Test type: Superiority; p = .28, t-test, 2 sided; df = 48
Statistical Analysis 3: Comparison: Typically Developing Children Immediate Intervention vs Down Syndrome Participants Immediate Intervention; Null Hypothesis: Amount of change in Perspective Taking will not differ for participants with Down Syndrome in the Immediate Intervention Condition who received16 weeks of experiential intervention and Typically Developing Children in the Immediate Intervention who also received 16 weeks of intervention; Test type: Superiority; p = .23, t-test, 2 sided; df = 55

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for approximately 18 weeks per individual. The time ranged from Baseline Data Collection (first session with each participant) until Final Outcome Data collection (last session with each participant), with Final Outcome Data Collection occurred following the16 weeks of experience training. Slight variations were possible when participants missed or rescheduled experience training over the 16-week period.
Description: No Down Syndrome participants were included in the Down Syndrome Participant Delayed condition. Hence, number of participants at risk for all categories of adverse event is this condition is identified as 0
Groups:
- Typically Developing Children Immediate Intervention: Child Participants received 16 weeks of spatial ability experience.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Typically Developing Children Deleayed Intervention: Child Participants received 8 weeks of spatial ability experience. Experience training was initiated eight weeks following the initial assessment (no intervening task) and immediately following the second assessment.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
- Down Syndrome Participants Intervention: Down Syndrome Participants received 8 weeks of spatial ability experience. Experience training was initiated eight weeks following the initial assessment (no intervening task) and immediately following the second assessment.
  Spatial Ability Experience: Participants will engage in puzzle construction, block play, visual search, hide and seek
Arm/Group | Typically Developing Children Immediate Intervention | Typically Developing Children Deleayed Intervention | Down Syndrome Participants Immediate Intervention | Down Syndrome Participants Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/24 | 0/30 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/24 | 0/30 | 0/0
Other Adverse Events (participants affected / at risk) | 0/30 | 0/24 | 0/30 | 0/0

LIMITATIONS AND CAVEATS:
Remote training due to CoVid increased duration of the project (16 instead of 8 weeks), made it difficult to recruit participants with Down Syndrome for the Delayed intervention condition. Hence, there is a need to modify the basic Data Analysis Plan, including using covariation procedures to account for difficulties matching groups. Still, the comparisons have yielded important results relevant to using experiential training to improve spatial abilities of individuals with Down Syndrome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT05332912/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT05332912/ICF_001.pdf